CLINICAL TRIAL: NCT00653016
Title: An Open Label Multicentre Study to Evaluate Patient Satisfaction and Preference for the EVRA Transdermal Contraceptive System Compared to Previously Used Contraceptive Method.
Brief Title: An Open-label, Multicentre Study on Preference and Satisfaction of Canadian Women for the Transdermal Contraceptive Patch vs. Previous Primary Contraceptive Method
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002908
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2010-03

CONDITIONS: Female Contraception
Keywords: Contraception; norelgestromin; ethinyl estradiol; transdermal contraceptive patch; EVRA; ORTHO EVRA
MeSH Terms: interventions — norelgestromin; Ethinyl Estradiol

INTERVENTIONS:
Drug: norelgestromin; ethinyl estradiol

SUMMARY:
The purpose of this study is to document the experience of transdermal contraceptive patch over a period of 9 cycles, compared to their previous contraceptive method.

DETAILED DESCRIPTION:
This was a multicentre, single-arm, open-label study. The objective of this phase IV study was to document the experience of women with the transdermal contraceptive patch (a weekly contraceptive patch delivering 150 mg norelgestromin/20 mg ethinyl estradiol daily) over a period of 9 cycles, compared to their previous contraceptive method. An open-label, multicentre, descriptive cohort study of 392 women requiring contraception were enrolled to receive the patch for nine cycles. A single treatment cycle consisted of three consecutive 7-day patch applications followed by one patch-free week. At the final visit, overall satisfaction and preference for the patch was rated compared to the previous contraceptive method.) The primary outcomes were treatment preference and overall satisfaction. Compliance, contraceptive efficacy, adhesion, and safety measures were secondary outcomes. Study participants were scheduled to receive the contraceptive patch for up to nine consecutive treatment cycles. Participants attended the clinic for 3 study visits: baseline/screening, Day 28 of Cycle 3 and Day 28 of Cycle 9 (or at early termination). A telephone interview was conducted on Day 28 of Cycle 6. Approximately 400 women were to be enrolled into the study and receive the transdermal contraceptive patch. Patients were recruited using ethics approved advertisements, in addition to investigators approaching patients presenting for routine well-woman checks. Participants who met all of the eligibility criteria were instructed to apply the first patch on the first day of their next menses (or 13 weeks following the last medroxyprogesterone acetate injection) and to wear this patch for seven days. They were then instructed to apply a new patch for weeks 2 and 3, and then be patch-free for week 4. Applying a new patch on the day after week 4 ended started a new cycle. All patches were to be applied/changed on the same day of the week and at approximately the same time of day. Only one patch was to be worn at a time. Patches could be applied to the buttocks, abdomen, upper outer arm, or upper torso (excluding breasts) and participants were instructed to apply new patches to a different site. Patches were to adhere on their own; no supplemental tape or adhesive was permitted. If a patch partially detached, participants could reapply it; however, patches that completely detached were to be replaced immediately and the replacement patch would be worn for the remainder of that week. Eligible patients were instructed to apply the 1st patch on the first day of their next menses (or 13 weeks following last medroxyprogesterone acetate injection) and to wear this patch for 7days. They were then instructed to apply a new patch for weeks 2 and 3, and then be patch-free for week 4. Applying a new patch on the day after week 4 ended started a new cycle. All patches were to be applied/changed on the same day of the week and at approximately the same time of day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females, who were sexually active and at risk of pregnancy were eligible to participate in this study provided that they had regular menses occurring every 25 to 35 days (except for those women using medroxyprogesterone acetate)
* women who were using one of the following methods of contraception as their primary method in the 3 months prior to admission: oral contraceptive, intrauterine device, medroxyprogesterone acetate injection, double-barrier method consisting of condoms and spermicidal foam or gel, or a diaphragm and spermicidal foam or gel
* study participants had to have a normal Pap smear within the previous 12 months
* a negative urine pregnancy test at admission
* have a systolic/diastolic blood pressure <= 140/90 mm Hg
* be within 35% of acceptable body mass index (upper limit of 32.4)
* be willing to switch their current method of contraception
* and agree not to use any other steroid hormonal therapy other than topical corticosteroids or inhaled corticosteroids for asthma, during the course of the study.

Exclusion Criteria:

* History or presence of disorders commonly accepted as contraindications to steroid hormonal therapy, e.g., deep vein thrombophlebitis, thromboembolic disorders, cerebral vascular or coronary artery disease, etc.
* Additionally, participants who were menopausal
* had skin conditions resulting in oily, irritated or damaged skin at all potential application sites
* Had a history or presence of dermal hypersensitivity
* The presently used contraceptive method were any of condoms alone, abstinence, withdrawal, or a rhythm method
* Had received medroxyprogesterone acetate injection <=12 weeks prior to enrolment
* had a history of alcohol or substance abuse within 12 months of enrolment
* had received any experimental drug or device within 30 days of enrolment
* Had used barbiturates, antiepileptics, rifampin, griseofulvin, or other hepatic enzyme inducing drugs within 30 days of enrolment
* Chronic systemic antibiotic use
* Had an uncontrolled thyroid disorder
* Were smokers over the age of 35
* Had Pap smear evidence of atypical squamous cells or adenocarcinoma or other malignancy
* Had a desire to conceive in the subsequent 9 months of enrolment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 405 (Actual)
Dates: Start 2002-10; Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Final visit - preference for patch vs. previous method, identify main reason for preference; satisfaction questionnaire with the previous contraceptive method at baseline and with the patch at the end of cycles 3, 6, 9 or early termination

SECONDARY OUTCOMES:
ongoing compliance based on dosing data recorded in diary cards; efficacy using the Pearl Index; patch adhesion using diary cards; adverse events at each visit, vital signs, body weigh changes, physical and gynaecological exams

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho Inc. Clinical Trial, Study Director — Janssen-Ortho Inc., Canada

REFERENCES:
- [Result] Weisberg F, Bouchard C, Moreau M, Audet MC, Mawdsley S, Dattani D, Dinniwell J, Horbay GL; NRGEEP-CON-401 Study Group. Preference for and satisfaction of Canadian women with the transdermal contraceptive patch versus previous contraceptive method: an open-label, multicentre study. J Obstet Gynaecol Can. 2005 Apr;27(4):350-9. doi: 10.1016/s1701-2163(16)30462-5. PMID 15937609